CLINICAL TRIAL: NCT02548624
Title: An Assessment of the Zephyr BioPatch and Its Ability to Monitor Patient Position
Status: Withdrawn | Type: Observational
Why Stopped: Protocol is being reevaluated by sponsor
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPO0520
Record Dates: First submitted 2015-09-01; First posted 2015-09-14 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Patient Positioning; Monitoring, Physiologic; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Zephyr BioPatch — The ZephyrLIFE Hospital System includes the BioPatch™ device (consisting of the BioModule™ sensor, BioModule™ holder, and snap ECG electrodes), the ECHO radio system, and a software monitoring interface. The BioModule™ sensor is a Class II device, 510(k) cleared by the FDA, and commercially available.
  The ZephyrLIFE Hospital System stores, transmits and displays vital sign data including ECG, HR, RR, body orientation, and activity to caregivers via a central station.
  Other Names: ZephyrLIFE Hospital System

SUMMARY:
The primary objective of the study is to examine the effectiveness of the Zephyr BioPatch in measuring position changes of a non-patient subject in a lab setting and to examine the effectiveness of the Zephyr BioPatch in measuring position changes of hospitalized patients.

ELIGIBILITY:
Inclusion Criteria for Laboratory Subject:

1. Signed and dated informed consent by subject
2. Male or female of any race
3. At least 18 years of age
4. Willingness to have study device attached during study participation
5. Willingness to participate in all aspects of the study

Exclusion Criteria for Laboratory Subject:

1. Implanted pacemaker or defibrillator
2. Allergy or sensitivity to ECG leads or similar types of adhesive
3. History of hospital admission or a surgical procedure in the 60 days prior to study enrollment
4. BMI > 30.0

Inclusion Criteria for Hospital Subjects:

1. Signed and dated informed consent by subject
2. Male or female of any race
3. At least 18 years of age
4. Expected hospitalized admission on the general care floor for at least three days
5. At risk for hospital-acquired pressure ulcers as defined by score on the Braden Scale of < 18
6. Willingness to have study devices attached during study participation
7. Willingness to participate in all aspects of the study

Exclusion Criteria for Hospital Subjects:

1. Implanted pacemaker or defibrillator
2. Allergy or sensitivity to ECG leads or similar types of adhesive
3. Subject will be sleeping in a chair or spending the majority of time in a chair
4. BMI > 39.9

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The laboratory observation will consist of one non-patient subject (N=1). The hospital observation will consist of 18 patients (N=18) hospitalized at the Columbia University Medical Center on the general care floor at-risk for hospital-acquired pressure ulcers. The hospitalized subjects will be stratified into three groups. Six subjects with normal BMI classification (18.5 -24.9), six with overweight BMI classification (25.0-29.9), and six with overweight BMI classification (30.0-39.9) will comprise the study sample.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Body position | During a 2.5 hour lab observation
  Body position will be classified as facing right, facing left, facing down (prone), or facing up (supine).
Body position | During a 24 hospital observation
  Body position when lying horizontally will be classified as facing right, facing left, facing down (prone), or facing up (supine).

SECONDARY OUTCOMES:
Performance of the Zephyr BioPatch position output in hospitalized patients of varying body mass indexes (BMI) | During a 24 hospital observation.
  Body position when lying horizontally will be classified as facing right, facing left, facing down (prone), or facing up (supine).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Adelman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States